CLINICAL TRIAL: NCT01449357
Title: A Single-arm Phase II Trial Investigating the Efficacy and Safety of Zalutumumab in Patients With Non-Small Cell Lung Cancer Who Have Progressive Disease After Treatment With Tyrosine Kinase Inhibitors
Brief Title: Zalutumumab in Non-Small Cell Lung Cancer (NSCLC) Patients Refractory to Tyrosine Kinase Inhibitors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial never initiated
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEN210
Record Dates: First submitted 2011-09-29; First posted 2011-10-10 (Estimated); Last update posted 2011-10-10 (Estimated); Status verified 2011-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; Zalutumumab; Efficacy; Safety
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — zalutumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- zalutumumab (Experimental)
  Interventions: Drug: zalutumumab

INTERVENTIONS:
Drug: zalutumumab — IV infusion, 16mg/kg on weekly basis until DP

SUMMARY:
A Single-arm Phase II Trial Investigating the Efficacy and Safety of Zalutumumab in Patients with Non-Small Cell Lung Cancer who have Progressive Disease after Treatment with Tyrosine Kinase Inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have documented disease progression after TKI treatment (verified by CT scan and/or MRI according to RECIST).

Exclusion Criteria:

* Estimated life expectancy of less than 3 months.
* Received the following treatments within 2 weeks prior to Visit 2:

  * Cytotoxic or cytostatic anti-cancer chemotherapy
  * Total resection or irradiation of the target lesion
  * Any investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Objective Response (OR) defined as complete response (CR) or partial response (PR) according to the RECIST criteria (revised version 1.1) within 6 months. | within 6 months

SECONDARY OUTCOMES:
Disease Control defined as CR, PR or Stable Disease (SD) according to the RECIST criteria (revised version 1.1) within 6 months. | within 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Not applicable, Study cancelled, Study Chair — H. Lee Moffitt Cancer Center, Tampa, Florida, USA